CLINICAL TRIAL: NCT04197063
Title: Evaluating a Portion Cap Policy on Sugar-Sweetened Beverages
Brief Title: Sugar-Sweetened Beverage Portion Limit Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Pamela Rothpletz-Puglia, EdD, RD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2019001933
Record Dates: First submitted 2019-10-10; First posted 2019-12-12 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Health Policy
Keywords: sweetened beverage; portion size; policy

STUDY DESIGN:
Intervention Model Description: This study randomized participants to one of four conditions: 1) Current SSB restaurant portion sizes with the option to purchase beverage refills; 2) Current SSB restaurant portions plus free refills; 3) </= 16 oz. SSB portions with the option to purchase beverage refills; or 4) </= 16 oz. SSB portions plus free refills.
Who Masked: Participant
Masking Description: The data was collected during a sham focus group where the purpose of the study was concealed from the participants. The purpose of the study was unmasked to participants when they returned on the following day and completed the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Current SSB restaurant portions purchase refill (Experimental): Offered a menu with current SSB restaurant portion sizes with the option to purchase refills
  Interventions: Behavioral: Sweetened beverage portion size limit
- Current SSB restaurant portions free refill (Experimental): Offered a menu with current SSB restaurant portion sizes plus free beverage refills
  Interventions: Behavioral: Sweetened beverage portion size limit
- </= 16 oz. SSB portions with the option to purchase refills (Experimental): Offered a menu with </= 16 oz. SSB portion sizes with the option to purchase refills
  Interventions: Behavioral: Sweetened beverage portion size limit
- </= 16 oz. SSB portions plus free refills (Experimental): Offered a menu with </= 16 oz. SSB portion sizes plus free refills
  Interventions: Behavioral: Sweetened beverage portion size limit

INTERVENTIONS:
Behavioral: Sweetened beverage portion size limit

SUMMARY:
This present study is an evaluation of de-identified data collected previously during a randomized controlled study (RCT). The objective of the original RCT titled "Sugar-Sweetened Beverage (SSB) Portion Limit Dining Lab RCT" was to examine the impact of limiting the portion size of SSB to 16 oz in a laboratory dining setting. The RCT was designed to assess the impact of limiting the size of SSB offered on a restaurant menu and the availability of free fills on beverage and food purchases, consumption and caloric intake at the test meal and subsequent meals (over a 24-hour period).

DETAILED DESCRIPTION:
Briefly, the data for this evaluation were collected from adults recruited from the Boston / Cambridge area to participate in an RCT conducted at an eating behavior lab at the Landmark Center (Lab). Participants were masked to the purpose of the study and were randomized to one of four conditions. To conceal the purpose of the study, participants were asked to participate in a pseudo-focus group pretending to conduct consumer research on restaurant preferences. Participants were asked not to eat after 3 pm prior to the 5:30 pm focus group. Participants were seated at individual dining tables and were asked to order and purchase dinner from a restaurant menu and consumed the meal while in the restaurant Lab. After the focus group, participants completed electronic questionnaires (e.g., demographic information, eating behaviors, and perceptions of the meal). Participants returned to the Lab the following day to complete a brief dietary recall interview. After they completed the study procedures, they were debriefed about the purpose of the study and provided the opportunity to withdraw from the study.

The current evaluation will be conducted under an IRB-approved, apriori, statistical analysis plan using the data collected during the Sugar-Sweetened Beverage (SSB) Portion limit Dining Lab RCT.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older
* Ability to speak and read English
* Willing to participate and follow protocol specified activities

Exclusion Criteria:

-Severe food allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2015-08-27 (Actual); Study Completion 2015-08-27 (Actual)

PRIMARY OUTCOMES:
Total calories food and beverages ordered from the study restaurant menu at the test dinner meal | Immediately after Day 1 test dinner meal
  Total calories ordered will be computed by summing the calories of each menu item selected for the test dinner meal.
  The calorie content for all food and drinks will be based on the nutritional information, posted on the restaurant's website for each menu item.
Total calories from food and drink consumed during the test the dinner meal | 24-hours post-Day 1 test dinner meal
  Calories consumed will be measured by weighing all food items before and after the test dinner meal using a digital scale accurate up to +0.1 grams. The weight of each plate/cup collected after the meal will be subtracted from the weight of each plate/cup prior to being served. The weight of the food in conjunction with the caloric density of each item will be combined to calculate the total caloric intake for each participant at the test dinner meal.

SECONDARY OUTCOMES:
Total beverage calories ordered at the dinner meal | Immediately after Day 1 test dinner meal
  The beverages calorie content of beverage items was based on the nutritional information available online.
Total beverage calories consumed at the dinner meal | Immediately after Day 1 test dinner meal
  Beverages were weighed before and after the meal to allow for the calculation of total beverage calories consumed. The calorie content of the beverage items was based on the nutritional information available online.
Total food calories ordered at the dinner meal | Immediately after Day 1 test dinner meal
  The food calorie content was based on the nutritional information available online.
Total food calories consumed at the dinner meal | Immediately after Day 1 test dinner meal
  Food items were weighed before and after the meal to allow for the calculation of total calories consumed. The calorie content of food items was based on the nutritional information available online.
Total calories consumed after the dinner meal | 24-hours post-Day 1 test dinner meal
  Total calories participants consumed after the dinner meal were measured with the National Cancer Institute's web-based Automated Self Administered 24-hour Dietary Recall program
Combination of calories consumed at dinner & post-dinner | From immediately after Day 1 test dinner meal until 24-hours post Day 1 dinner meal
  This will be calculated by adding the value for total calories consumed at the dinner meal to the value for total calories consumed post-dinner.

OTHER OUTCOMES:
Overall satisfaction with the price of the food item/s ordered: 7-point Likert item | Immediately after Day 1 test dinner meal
  7-point Likert item (1= not at all satisfied; 7= extremely satisfied]
Overall satisfaction with the portion of the food item/s ordered: 7-point Likert item | Immediately after Day 1 test dinner meal
  7-point Likert item (1= not at all satisfied; 7= extremely satisfied]
Satisfaction with drink size | Immediately after Day 1 test dinner meal
  Too small, Just right, Too big
Pre-meal hunger | Immediately after Day 1 test dinner meal
  Before eating this meal, how hungry were you? [7-point Likert item (1= not at all hungry, 7= extremely hungry)]

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Roberto, PhD, Study Director — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data will be made publically available, upon request
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data and supporting information will become available starting 6 months after the final analysis is completed and the summary data are published.
Access Criteria: Contact the Study Investigators for information on how to access the data and supporting information